CLINICAL TRIAL: NCT04790851
Title: A Randomized, Controlled, Multicenter Phase 4 Clinic Trial to Evaluate the Immunogenicity and Safety of Combined Immunization of Inactivated SARS-CoV-2 Vaccines (Vero Cell) (COVAX) (Produced in Beijing) and 23-valent Pneumococcal Polysaccharide Vaccine (PPV23) or Quadrivalent Inactivated Influenza Vaccine (IIV4)
Brief Title: Evaluation of Immunogenicity and Safety of Combined Immunization of COVID-19 Vaccine (Produced in Beijing) and PPV23 / IIV4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Chengdu Institute of Biological Products Co.,Ltd. (Industry); Changchun Institute of Biological Products Co., Ltd. (Industry); Beijing Institute of Biological Products Co Ltd. (Industry); Sichuan Center for Disease Control and Prevention (Other Government); Shanghai Municipal Center for Disease Control and Prevention (Other); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COVAX+PPV23+IIV4-Beijing
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Influenza, Human; Pneumonia, Pneumococcal; Covid19
MeSH Terms: conditions — Influenza, Human; Pneumonia, Pneumococcal; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: serum testing technicians were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Experimental Group (384 subjects) will receive: 1st dose : combined vaccination of COVAX+IIV4; 2nd dose: combined vaccination of COVAX+PPV23
  Interventions: Biological: COVAX+IIV4; COVAX+PPV23
- Control group A (Active Comparator): Control Group A (384 subjects) will receive: 1st dose: COVAX only; 2nd dose: COVAX only
  Interventions: Biological: COVAX only (1st and 2nd dose)
- Control group B (Active Comparator): Control Group B (384 subjects) will receive: 1st dose: IIV4 only; 2nd dose: PPV23 only
  Interventions: Biological: IIV4 for the 1st dose and PPV23 for the 2nd dose

INTERVENTIONS:
Biological: COVAX+IIV4; COVAX+PPV23 — 1st dose : combined vaccination of COVAX+IIV4; 2nd dose: combined vaccination of COVAX+PPV23
  Arms: Experimental group
Biological: COVAX only (1st and 2nd dose) — 1st dose: COVAX only; 2nd dose: COVAX only
  Arms: Control group A
Biological: IIV4 for the 1st dose and PPV23 for the 2nd dose — 1st dose: IIV4 only; 2nd dose: PPV23 only
  Arms: Control group B

SUMMARY:
Subjects will be recruited and divided into 3 groups:

Experimental Group (384 subjects): 1st dose : combined vaccination of COVAX+IIV4, 2nd dose: combined vaccination of COVAX+PPV23; Control Group A (384 subjects): 1st dose: COVAX only, 2nd dose: COVAX only; Control Group B (384 subjects): 1st dose: IIV4 only, 2nd dose: PPV23 only.

Blood samples will be collected 3 times:

before the 1st dose of vaccinatioin; before the 2nd dose of vaccination; 28 days after the 2nd dose of vaccination.

The immunogenicity and safety of both experimental and control groups will be analyzed.

DETAILED DESCRIPTION:
This randomized, parallel, controlled study is designed to evaluate the immunogenicity and safety of simultaneously immunization of COVAX + PPV23 and COVAX + IIV4.

1152 subjects are divided into 3 groups, including 1 experimental group and 2 control groups (control group A and B). Each group includes 384 subjects respectively.

Experimental Group (384 subjects) will receive: 1st dose : combined vaccination of COVAX+IIV4, 2nd dose: combined vaccination of COVAX+PPV23; Control Group A (384 subjects) will receive: 1st dose: COVAX only, 2nd dose: COVAX only; Control Group B (384 subjects) will receive: 1st dose: IIV4 only, 2nd dose: PPV23 only.

Specifically, each group will be divided again. Each 384-subject group is divided again into 2 age-based subgroups: (1) 18-59 years old; (2) ≥60 years old.

Each subgroup includes 192 subjects respectively. Blood samples will be collected 3 times: (1) before the 1st dose of vaccinatioin; (2) before the 2nd dose of vaccination; (3) 28 days after the 2nd dose of vaccination.

To evaluate the immunogenicity, the investigators will detect and compare the neutralizing antibody levels, the seroconversion rates and antibody geometric mean concentrations.

The safety of all groups will be monitored as well.

ELIGIBILITY:
Inclusion criteria:

* ≥18 years old when enrolled;
* Participants signing the informed consent;
* Being able to participate in all planned follow-ups and accomplish all research procedures including completing a diary card and coming back for interview;
* Having not been administered any pneumonia vaccine or COVID-19 vaccine, and having not been administered an influenza vaccine in the current season before enrollment;
* ≥14 days from the most recent vaccination;
* Before enrollment, the body temperature is ≤37.0C as confirmed by medical history and clinical examination.

Exclusion criteria for the first dose:

* Having a history of COVID-19 or a positive nucleic acid test for COVID-19;
* Having a history or a family history of allergy, convulsion, epilepsy, brain disease, or mental illness;
* Being allergic to any component of vaccines, or having a history of severe allergic reaction to any vaccine;
* Having immunodeficiency disorder, during treatment of malignant tumor, having immunodeficiency induced by immunosuppressants (oral steroid hormones) or HIV, or having a family member with close contact who suffers from congenital immune disorder;
* Having injection of non-specific immunoglobulin within 1 month prior to enrollment;
* Having acute febrile illness or communicable disease;
* Having a history of confirmed thrombocytopenia or other coagulation disorders, which may cause contraindications for a subcutaneous injection;
* Having severe chronic disease or acute exacerbation of chronic disease, or having uncontrolled hypertension or diabetes;
* Having various infectious, pyogenic, or allergic skin diseases;
* Women in pregnancy or lactation or participants who plan for a baby within 3 months after vaccination should delay the vaccination;
* Having any condition that may affect trial assessment as determined by researchers.

Exclusion criteria for the second dose:

* Having any serious adverse event related to the first dose vaccination;
* After vaccination, having systemic adverse reaction or allergic reaction with a severity of grade 3 or higher as determined by researchers;
* Having a newly emerging condition that meets the exclusion criteria for the first dose;
* Having any condition that may affect trial assessment as determined by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1133 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate (COVAX) | Results obtained 28 days after the first dose (= right before the second dose)
  the rate of positive seroconversion against coronavirus
Seroconversion rate (COVAX) | Results obtained after the second dose of vaccination (= 56 days after the first dose, or 28 days after the second dose)
  the rate of positive seroconversion against coronavirus
Neutralizing antibody level (COVAX) | Baseline (before vaccination) results
  neutralizing antibody level against coronavirus
Neutralizing antibody level (COVAX) | Results obtained 28 days after the first dose (= right before the second dose)
  neutralizing antibody level against coronavirus
Neutralizing antibody level (COVAX) | Results obtained after the second dose of vaccination (= 56 days after the first dose, or 28 days after the second dose)
  neutralizing antibody level against coronavirus
Seropositive rate (IIV4) | Baseline (before vaccination) results
  the rate of positive seroconversion against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Seroconversion rate (IIV4) | Results obtained 28 days after the first dose (= right before the second dose)
  the rate of positive seroconversion against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Seroconversion rate (IIV4) | Results obtained after the second dose of vaccination (= 56 days after the first dose, or 28 days after the second dose)
  the rate of positive seroconversion against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Hemmagglution inhibition antibody level (IIV4) | Baseline (before vaccination) results
  Hemmagglution inhibition antibody levels against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Hemmagglution inhibition antibody level (IIV4) | Results obtained 28 days after the first dose (= right before the second dose)
  Hemmagglution inhibition antibody levels against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Hemmagglution inhibition antibody level (IIV4) | Results obtained after the second dose of vaccination (= 56 days after the first dose, or 28 days after the second dose)
  Hemmagglution inhibition antibody levels against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Seroconversion rate (PPV23) | Results obtained 28 days after the first dose (= right before the second dose)
  the rate of positive seroconversion against 23 pneumococcal serotypes
Seroconversion rate (PPV23) | Results obtained after the second dose of vaccination (= 56 days after the first dose, or 28 days after the second dose)
  the rate of positive seroconversion against 23 pneumococcal serotypes
Neutralizing antibody level (PPV23) | Baseline (before vaccination) results
  Neutralizing antibody level against 23 pneumococcal serotypes
Neutralizing antibody level (PPV23) | Results obtained 28 days after the first dose (= right before the second dose)
  Neutralizing antibody level against 23 pneumococcal serotypes
Neutralizing antibody level (PPV23) | Results obtained after the second dose of vaccination (= 56 days after the first dose, or 28 days after the second dose)
  Neutralizing antibody level against 23 pneumococcal serotypes

SECONDARY OUTCOMES:
Adverse events following vaccination | 0-6 months
  analyse the incidence of adverse events following immunization, both solicited and unsolicited

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, Principal Investigator — Shanghai Municipal Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Sichuan Center for Disease Control and Prevention, Chengdu
  - Shanghai Municipal Center for Disease Control and Prevention, Shanghai
  - Shanxi Provincial Center for Disease Control and Prevention, Taiyuan

REFERENCES:
- [Derived] Chen H, Huang Z, Chang S, Hu M, Lu Q, Zhang Y, Wang H, Xiao Y, Wang H, Ge Y, Zou Y, Cui F, Han S, Zhang M, Wang S, Zhu X, Zhang B, Li Z, Ren J, Chen X, Ma R, Zhang L, Guo X, Luo L, Sun X, Yang X. Immunogenicity and safety of an inactivated SARS-CoV-2 vaccine (Sinopharm BBIBP-CorV) coadministered with quadrivalent split-virion inactivated influenza vaccine and 23-valent pneumococcal polysaccharide vaccine in China: A multicentre, non-inferiority, open-label, randomised, controlled, phase 4 trial. Vaccine. 2022 Aug 26;40(36):5322-5332. doi: 10.1016/j.vaccine.2022.07.033. Epub 2022 Jul 29. PMID 35931636